CLINICAL TRIAL: NCT02011672
Title: Effect of Milk Ingredients on Glucose Regulation and Inflammation in Overweight Subjects
Brief Title: Effect of Milk Ingredients on Glucose Regulation and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Alwine Kardinaal, Project Manager Health, NIZO Food Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL46103.081.13
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Glucose Regulation; Low-grade Inflammation
Keywords: dairy; glucose; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nutrient-enriched milk (Experimental): consumption of 250 ml three times per day
  Interventions: Other: nutrient-enriched milk
- regular milk (Placebo Comparator): consumption of 250 ml three times per day
  Interventions: Other: regular milk

INTERVENTIONS:
Other: nutrient-enriched milk
  Arms: nutrient-enriched milk
Other: regular milk
  Arms: regular milk

SUMMARY:
Background: Recent advances in science have established a fundamental role for low grade chronic inflammation in mediating all stages of most of the non-communicable diseases associated with ageing. Pro-inflammatory effects of hyperglycemia have been described. Dairy and its components are known to exert beneficial effects on postprandial hyperglycemia. This study investigates if dairy, normal and enriched, can reduce chronic inflammation via improvement in glucose regulation.

Objective: To compare the effect of a nutrient-enriched dairy drink on parameters of glucose regulation and postprandial inflammation with the effect of a standard milk drink, within a population of overweight, apparently healthy subjects.

Study design: The study is designed as a double-blind randomized placebo-controlled parallel trial during 7 weeks, during which the test and reference products will be consumed at home.

Main study parameters/endpoints: The difference in absolute change in fasting blood plasma concentration of glucose, insulin and IL-6, from baseline to endpoint, and the difference in postprandial response of plasma concentration of glucose, insulin and IL-6 at the end of the treatment period, between subjects consuming the test and reference product.

ELIGIBILITY:
Inclusion Criteria:

* BMI 28-35 kg/m2
* Waist circumference >102 cm
* Healthy as assessed by the NIZO lifestyle and health questionnaire and results of the pre-study safety laboratory tests.
* Regular and normal Dutch eating habits as assessed by the NIZO lifestyle and health questionnaire (3 main meals per day)
* Habitual consumption of dairy products as assessed by dietary questionnaire
* Voluntary participation
* Having given written informed consent
* Willing to comply with study procedures
* Access to internet
* Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data for at least 15 years.
* Willing to accept disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
* Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous or inhalatory administration of substances
* Having a history of medical or surgical events that may significantly affect the study outcome, including: Inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding; major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; known or suspected gastrointestinal strictures
* Medical drug use; antibiotics, laxatives, glucose lowering drugs, insulin; all medication with an inflammation inhibiting effect (e.g. NSAIDS, corticosteroids) and/or an effect on blood coagulation (e.g. coumarins, inhibitors of thrombin or factor Xa, acetylsalicylic acid, antidepressants from the group of serotonin reabsorption inhibitors, tranexamin acid)
* Mental status that is incompatible with the proper conduct of the study
* A self-reported reported food allergy or sensitivity (wheat, milk, lactose, eggs, nuts, etc)
* Alcohol consumption > 28 units/week and 4/day
* Exercise > 3 hours/week
* Smoking >20 cigarettes/day
* Reported unexplained weight loss or weight gain of > 3 kg in the month prior to pre-study screening
* Reported slimming or medically prescribed diet
* Reported vegan or macrobiotic life-style
* Recent blood donation (<1 month prior to Day 01 of the study)
* Not willing or afraid to give up blood donation during the study
* Personnel of NIZO food research or Wageningen University, department of Human Nutrition, their partner and their first and second degree relatives
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
change in fasting blood glucose | baseline and 7 weeks
change in fasting plasma interleukin-6 (IL-6) | baseline and 7 weeks

SECONDARY OUTCOMES:
postprandial area under the curve for plasma glucose | 7 weeks
change in fasting insulin | 7 weeks
postprandial area under the curve for plasma insulin | 7 weeks
postprandial area under the curve for plasma IL-6 | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alwine Kardinaal, PhD, Principal Investigator — NIZO Food Research
Locations (1):
- NIZO food research, Ede, Netherlands